CLINICAL TRIAL: NCT00365768
Title: A Pilot Study Investigating the Effects of Glutamine and Vincristine-Induced Neuropathy in Pediatric Patients With Cancer
Brief Title: Glutamine in Treating Neuropathy Caused by Vincristine in Young Patients With Lymphoma, Leukemia, or Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Julia Glade Bender, Irving Assistant Professor of Clinical Pediatrics, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AAAA6806; CPMC-ICCR-3349 (Other: Columbia University Medical Center)
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Results first posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-07

CONDITIONS: Kidney Cancer; Leukemia; Lymphoma; Neurotoxicity; Peripheral Neuropathy; Sarcoma
Keywords: stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage II childhood small noncleaved cell lymphoma; stage I Wilms tumor; stage II Wilms tumor; stage III Wilms tumor; stage IV Wilms tumor; stage V Wilms tumor; childhood grade III lymphomatoid granulomatosis; childhood diffuse large cell lymphoma; childhood immunoblastic large cell lymphoma; stage I childhood large cell lymphoma; stage I childhood lymphoblastic lymphoma; stage I childhood small noncleaved cell lymphoma; stage II childhood large cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood large cell lymphoma; stage IV childhood lymphoblastic lymphoma; stage IV childhood small noncleaved cell lymphoma; childhood Burkitt lymphoma; stage III childhood small noncleaved cell lymphoma; untreated childhood acute lymphoblastic leukemia; childhood nasal type extranodal NK/T-cell lymphoma; previously untreated childhood rhabdomyosarcoma; localized Ewing sarcoma/PNET; metastatic Ewing sarcoma/PNET; neurotoxicity; peripheral neuropathy
MeSH Terms: conditions — Kidney Neoplasms; Leukemia; Lymphoma; Neurotoxicity Syndromes; Peripheral Nervous System Diseases; Sarcoma; Burkitt Lymphoma; Wilms Tumor; Lymphoma, Large B-Cell, Diffuse; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Extranodal NK-T-Cell; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Glutamine; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: Glutamine (Experimental): Beginning 1 week after administration of vincristine chemotherapy, patients receive oral glutamine twice daily on days 1-21.
  Interventions: Drug: Glutamine
- Arm II: Placebo (Placebo Comparator): Beginning 1 week after administration of vincristine chemotherapy, patients receive oral placebo twice daily on days 1-21.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Glutamine — Administered orally twice daily for 21 days
  Other Names: Nutritional Supplement
  Arms: Arm I: Glutamine
Other: Placebo — Administered orally twice daily for 21 days
  Arms: Arm II: Placebo

SUMMARY:
RATIONALE: Glutamine may help lessen neuropathy caused by chemotherapy. It is not yet known whether glutamine is more effective than a placebo in treating neuropathy caused by vincristine.

PURPOSE: This randomized phase II trial is studying glutamine to see how well it works compared to a placebo in treating neuropathy caused by vincristine in young patients with lymphoma, leukemia, or solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the incidence of vincristine-induced peripheral neuropathy in pediatric patients with lymphoma, leukemia, or solid tumors.

Secondary

* Compare the safety of glutamine vs placebo in these patients.
* Compare the efficacy of glutamine vs placebo in reducing the progression and/or resolution of vincristine-induced peripheral neuropathy in these patients.
* Compare the effect of glutamine supplementation vs placebo on chemotherapy-related toxicities in these patients.
* Compare the effect of glutamine vs placebo on measures of quality of life in these patients.
* Compare the effect of glutamine supplementation vs placebo on serum nerve growth factor and glutamine levels in these patients.
* Determine the effect of glutamine on vincristine-mediated antitumor efficacy in vitro.

OUTLINE: This is a randomized, double-blind, placebo-controlled, pilot study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Beginning 1 week after administration of vincristine chemotherapy, patients receive oral glutamine twice daily on days 1-21.
* Arm II: Beginning 1 week after administration of vincristine chemotherapy, patients receive oral placebo twice daily on days 1-21.

Patients in both arms undergo neuropsychological and clinical neurological assessment, blood collection for serum marker (e.g., serum glutamine and nerve growth factor) analysis, and quality of life assessment on days 1, 21, and 42.

After completion of study treatment, patients are followed for an additional 21 days.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the age of 5 and 21 years old.
* Patients who demonstrate the ability to complete the assessment instruments at baseline.
* Patients who are diagnosed with leukemia or solid tumors and are expected to receive a cumulative dose of > or = to 6mg/m2 of vincristine, or > 6mg if individual vincristine doses are capped at 2mg according to primary cancer treatment protocol, over a 30-week period.

Exclusion Criteria:

* Patients with primary CNS tumors other than medulloblastoma or patients with CNS metastasis.
* Patients with recurrent disease.
* Patients with Grade II, III or IV neurological status by the NCI CTC (Ver. 3.0) on clinical exam.
* Patients who have already received > 8mg/m2 of vincristine, or > 8mg if individual vincristine doses are capped at 2mg according to primary cancer treatment protocol, during their course of therapy at time of consent.
* Patients with hepatic encephalopathy or hyperammonemia.
* Patients with a focally abnormal neurologic exam.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2004-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia L. Glade-Bender, MD, Principal Investigator — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were consented according to Institutional Review Board approved guidelines during out routine outpatient or inpatient stay. The period of recruitment was from January 2007 to July 2011.
Pre-assignment Details: Fifty-six patients were enrolled and 49 were evaluable, with the reasons for removal from study after randomization due to: change in clinical status (N=3), family withdrew (N=2), family relocation (N=1) and other (N=1). 49 patients were randomized to the glutamine or placebo arm.
Period: Overall Study
Arm/Group | Arm I: Glutamine | Arm II: Placebo
Started | 24 | 25
Completed | 24 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Fifty-six patients were enrolled and 49 were evaluable.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Glutamine | Arm II: Placebo | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Continuous [Median (Full Range); unit: years] | 11 [5 to 19] | 10 [4 to 17] | 11 [4 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 10 | 13 | 23
Region of Enrollment [Number; unit: participants]
  United States | 24 | 25 | 49

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Vincristine-induced Peripheral Neuropathy
Time Frame: Up to 30 weeks from baseline while on Vincristine treatment
Measure: Number; unit: participants
Arm/Group | Arm I: Glutamine | Arm II: Placebo
Number analyzed (Participants) | 24 | 25
participants | 24 | 25

2. Secondary Outcome: Number of Participants With Progression of Neuropathy
Time Frame: 42 days
Measure: Number; unit: participants
Arm/Group | Arm I: Glutamine | Arm II: Placebo
Number analyzed (Participants) | 24 | 25
participants | 11 | 19

ADVERSE EVENTS:
Groups:
- Arm II: Beginning 1 week after administration of vincristine chemotherapy, patients receive oral placebo twice daily on days 1-21.
  Placebo: Administered orally twice daily for 21 days
Arm/Group | Arm I: Glutamine | Arm II
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 0/24 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes